CLINICAL TRIAL: NCT00227825
Title: Motivational Enhancement Therapy to Reduce Risk Behaviors in HIV Infected Youth
Brief Title: The Aim of This Study is to Determine the Effectiveness of a Motivational Enhancement Intervention in Reducing Risk Behaviors (Drug and Alcohol Use, Sexual Risk Behavior, Poor Adherence to Medications) Among HIV+ Youth. - 1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Wayne State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-14710-1; R21-14710-1
Record Dates: First submitted 2005-09-27; First posted 2005-09-28 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2005-09

CONDITIONS: Adherence; HIV Risk Behaviors; Alcohol & Drug Use; Health Behaviors; Sexual Risk Behaviors
Keywords: Behavioral Intervention
MeSH Terms: conditions — Substance-Related Disorders; Health Behavior | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Motivational interviewing

SUMMARY:
The purpose of this study is to conduct a pilot study of Motivational Enhancement Therapy (MET), an empirically validated behavioral change strategy, with young adults who are HIV +. The aim is to determine if MET is effective in increasing general health promotion behaviors, adherence to HIV+ specific medical treatment over and above taking medication, and decreasing risky behaviors in young adults who are HIV positive. The longer-term objective is to identify and way to decrease HIV transmission rates, disease progression, illness episodes, and hospitalizations in this high-risk population.

Hypotheses: 1)Youth receiving the motivational intervention plus referrals will report greater reductions in risky behaviors than youth in the control group receiving standard care plus referrals at 3-months post-baseline. This hypothesis will first be tested in the whole sample using an overall risk index. Then, the hypothesis will be tested with each behavior (reduced drug and alcohol use, condom use, taking medications,) within the subgroups reporting problem levels of that behavior; 2)Youth in the intervention group will demonstrate improved viral loads, will report greater improvement in perceived health status, depression, general psychological distress, disclosure to sexual partners, and will demonstrate greater attendance of medical and support service appointments than youth in the control group at 3 months post-baseline; 3)Youth in the intervention group will report greater reductions in temptation to engage in risky behaviors, increased self-efficacy, and improvements in readiness to change their behavior than youth in the control group at 3 months post-baseline; 4)The differences between the intervention and control group from pre- to post- intervention will be maintained at 6, 9, 12, and 15 months post-baseline (3, 6, 9, and 12 months after intervention completion).

DETAILED DESCRIPTION:
The proposed study is a randomized clinical trial with a wait-list control. The sample will be 60 HIV+ young adults between the ages of 16 to 24 years recruited from the DMC Horizons Project and other community based HIV programs. Self referred persons meeting the diagnostic criteria of HIV+ will also be accepted. There are no exclusion criteria. Subjects will be randomly assigned to one of 2 groups: MET NOW or MET LATER. MET LATER is the wait list control group. The only difference between the groups is the timing of the intervention and data collection. All subjects will complete 5 research visits and 4 MET therapy sessions. Research visits consists of an interview, completion of self-report questionnaires, a 20cc blood drawn for complete blood count (CBC), viral load and CD4 count, and adherence rating completed by the physician. Established questionnaires are used to measure health behaviors, sexual risk behaviors, substance use, self-efficacy, stage of change, social support, health beliefs, and mental health status. Research visits take about 1 = hours. Therapy sessions consist of MET provided by a trained therapist. Sessions last about 1 hour and focus on changing behavior to improve health, increase medical adherence, and/or reduce risk. Subjects choose the behaviors they want to change. There are a total of 4 sessions over 3 months. The MET NOW group will begin session immediately after the first (baseline) research visit and the MET LATER group will begin therapy sessions approximately 9 months after the first research visit. All subjects will be paid $25.00 for the first research visit with a $5 increase for each subsequent research visit, a total of $175.00 for the 5 research visits. Subjects will receive $10 gift certificate at each therapy session. Cab vouchers or parking fees will be provided for each therapy or research session.

ELIGIBILITY:
Inclusion Criteria:

* A sample of 60 HIV+youth, ages 16-24, will be recruited from the four health care sites in the Michigan Title IV Project.

Exclusion Criteria:

* In order to increase the likelihood that the current intervention will be easily transportable to real world settings, exclusion criteria are kept to a minimum. No exclusions will be made due to co-morbid mental health problems ( i.e. ADHD, conduct disorder, depression, anxiety disorder), with the exception of thought disorder (i.e. schizophrenia, autism). It is assumed that severe psychosis in conjunction with HIV may require management strategies beyond the scope of the MET interventions (i.e. residential placement). As resources are not available in the current grant to hire and train therapists who are bilingual or translate study questionnaires/measures, subjects will required to speak English fluently. Hispanic or Arabic families who meet this criterion will be included in the study. Currently, all clients at the clinic sites meet this last criterion.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 2002-01; Study Completion 2005-08

PRIMARY OUTCOMES:
Reduction of Risk Behaviors (Sexual, Drug, & Health), Viral Burden & CD4+ T Cell Count

SECONDARY OUTCOMES:
SES, health beliefs, physical and mental status, self-efficacy, stages of change, service utilization, HIV stigma

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Naar-King, Ph.D., Principal Investigator — Wayne State University
Locations (1):
- Detroit Medical Center-CHM and UHC, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No